CLINICAL TRIAL: NCT00828633
Title: Patient-Reported Outcomes For Gay Men With Localized Prostate Cancer
Brief Title: Health-Related Quality of Life in Gay Men With Localized Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Latini, Adjunct Assistant Professor of Urology, Baylor College of Medicine
Other Study IDs: CDR0000600597; BCM-H-21892 (Other: Baylor College of Medicine)
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Gathering information about prostate cancer, treatment, and quality of life from gay men with prostate cancer may help doctors plan the best treatment.

PURPOSE: This clinical trial is collecting information about health-related quality of life from gay men with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To enroll 200 gay men with localized prostate cancer in a cross-sectional study of prostate cancer outcomes.
* To complete an R01 application using pilot data collected from these patients.
* To complete manuscripts describing the factors that influence quality of life and treatment satisfaction in these patients.

OUTLINE: Patients complete a web-based survey about their disease (biopsy Gleason score, PSA at diagnosis, and T-stage), treatment (treatment type, time since treatment, and use of healthcare services [e.g., oral medications for erectile dysfunction]), symptom distress, and psychosocial factors (ethnicity, health literacy, level of social support, communication with provider, relationship status, and communication with partner) that affect their health-related quality of life. The data will be used to provide the information necessary to tailor an existing prostate cancer survivorship intervention to address the specific needs of gay men with prostate cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized prostate cancer

  * No advanced disease
* Self-identified as gay

PATIENT CHARACTERISTICS:

* Able to complete an online questionnaire
* Able to speak and understand English

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample contacted via Internet
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of disease factors and treatment factors on subjective well-being | Cross-sectional retrospective study, one timepoint
Effect of disease factors and treatment factors on illness intrusiveness | Cross-sectional retrospective study, one timepoint
Effect of psychosocial factors on subjective well-being | Cross-sectional retrospective study, one timepoint

CONTACTS AND LOCATIONS:
Overall Officials: David M. Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (2):
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
- Ryerson University, Toronto, Ontario, Canada